CLINICAL TRIAL: NCT05287282
Title: Impact of TECAR Therapy in Treatment of Post-natal Rectus Diastasis
Brief Title: Impact of TECAR in Treatment of Rectus Diastasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Rafat, Lecturer of physical therapy, Basic Sciences department, Physical therapy faculty, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT/WH
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Rectus Diastasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TECAR application (Experimental)
  Interventions: Other: TECAR application
- selected abdominal exercises program (Active Comparator)
  Interventions: Other: TECAR application

INTERVENTIONS:
Other: TECAR application — Radiofrequency (RF) is the emission of high frequency waves via an applicator. The transfer of electromagnetic energy stimulates targeted tissues. RF can be used in two ways: capacitive or resistive The capacitive mode (CET) concentrates the energy to target soft tissues containing electrolytes: muscles, vascular or lymphatic tissues. The resistive mode (RET) targets denser tissues containing more fat and fiber (such as bones, ligaments and tendons). High frequency waves penetrate deep into tissues and increase both exchanges and temperature and a recent study has demonstrated the effects of RF on the skin microcirculation and the intramuscular blood flow

SUMMARY:
The study aim to evaluate the impact of TECAR treatment on rectus diastasis in postnatal women

DETAILED DESCRIPTION:
Radiofrequency (RF) is the emission of high frequency waves via an applicator. The transfer of electromagnetic energy stimulates targeted tissues. RF can be used in two ways: capacitive or resistive ( Kumarane etal.,2015) This has been shown to increase vascularization and reduce inflammation and swelling and to accelerate the healing process and provide pain relief( Duñabeitia et al., 2018). It is used to provide rapid pain relief for sport injuries and allows quicker recovery [Duñabeitia etal, 2018& Weber T, Kabelka2011). low back pain and traumatology and urology (Notarnicola etal, 2017). The capacitive mode (CET) concentrates the energy to target soft tissues containing electrolytes: muscles, vascular or lymphatic tissues. The resistive mode (RET) targets denser tissues containing more fat and fiber (such as bones, ligaments and tendons). High frequency waves penetrate deep into tissues and increase both exchanges and temperature and a recent study has demonstrated the effects of RF on the skin microcirculation and the intramuscular blood flow (Kumaraane et al., 2015). To date, no study has evaluated the impact of TECAR treatment on rectus diastasis in postnatal women This study will be carried out on 30 postnatal females suffering from diastasis recti more than 2.5 cm with bulged abdomen, they will be selected from out patient physical therapy clinic, kafr el sheikh university. Their age ranged from 25 - 35 years. Their body mass index (BMI) ranged from 25-35 kg/m2. All women delivered normally

Exclusion criteria:

Any participant was excluded if she had any disease that interferes with exercises (asthma), any skin disease or sensitivity that interferes with the application, any chest disease or cardiac disease or women had abdominal or surgery.

All participants will read an explanation of the experimental procedures and sign an informed consent that is approved by the Ethical committee Institutional Review Board, Faculty of Physical Therapy, kafr elsheikh University, Egypt This study will be a randomized, double-blind, pre test-post test crossover trial with control group. The randomization procedure will be performed by a simple drawing of lots (A or B) which determined whether participants would receive the TECAR therapy and abdominal exercises ( group A) and abdominal exercises only in (group B). The randomization procedure will be performed through a computer program (Microsoft Excel 2010) that created a random table of numbers in which each number corresponded to the group A or B. After that, participants will be allocated according to the corresponding number of their allocation code. A researcher will be conducted the drawing procedures without informing participants and evaluators, to determine which will be in group A or group B. Thus, both participants and evaluators will be blinded to the allocation of treatment.

Study group (Group A):

It was consisted of 15 post natal women who will performed weight reduction diet ( 1200 kcal/day) , TECAR application and selected abdominal exercises program that consists of static abdominal and posterior pelvic tilting

Control group(Group B):

It was consisted of 15 postnatal women who was performed weight reduction diet (1200 kcal/day) and selected abdominal exercises and posterior pelvic tilting exercises.

ELIGIBILITY:
Inclusion Criteria:

* postnatal females suffering from diastasis recti more than 2.5 cm with bulged abdomen,
* Their age ranged from 25 - 35 years.
* Their body mass index (BMI) ranged from 25-35 kg/m2.
* All women delivered normally

Exclusion Criteria:

* Any participant was excluded if she had any disease that interferes with exercises (asthma), any skin disease or sensitivity that interferes with the application, any chest disease or cardiac disease or women had abdominal surgery.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
rectus abdominis cross section area | 1 cycle (42 days)
fat thickness | 1 cycle (42 days)
intra-recti distance | 1 cycle (42 days)

CONTACTS AND LOCATIONS:
Overall Officials: Eman A Elhosary, Professor, Principal Investigator — Assistant professor of physical therapy, Physical therapy faculty, Kafrelsheikh University
Locations (1):
- Kafrelshiesk university hospital, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No